CLINICAL TRIAL: NCT04283669
Title: Open-label, Phase 2 Clinical Trial of Crizotinib for Children and Adults With Neurofibromatosis Type 2 and Progressive Vestibular Schwannomas
Brief Title: Phase 2 Clinical Trial of Crizotinib for Children and Adults With Neurofibromatosis Type 2 and Progressive Vestibular Schwannomas
Acronym: NF110
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Girish Dhall, MD, Chair of of the NFCTC; Protocol PI, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300003645; W81XWH-17-2-0037 (Other Grant/Funding Number: CDMRP of the Dept. of Defense, US Army)
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Neurofibromatosis 2; Progressive Vestibular Schwannoma (VS)
MeSH Terms: conditions — Neurofibromatosis 2 | interventions — Crizotinib

STUDY DESIGN:
Intervention Model Description: Subjects with Neurofibromatosis Type 2 (NF2) and progressive vestibular schwannoma (VS) will be treated with crizotinib administered orally. Crizotinib will be taken continuously until disease progression or unacceptable toxicity, in continuous treatment cycles of 28 days each, for a maximum of 12 cycles. Clinical response will be assessed by MRI (volumetrics, primary objective) and audiology at the end of every 3rd cycle. Subjects with volumetric tumor progression will be taken off protocol. Patients who complete 12 cycles of treatment without disease progression, but within the following 24 weeks show subsequent disease progression (defined as >20% increase in target tumor volume compared to off-treatment volume), will be eligible for re-treatment on study for up to 48 additional weeks, provided they still meet study eligibility criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Continuous Treatment (Other): Subjects with Neurofibromatosis Type 2 (NF2) and progressive vestibular schwannoma (VS) will be treated with crizotinib administered orally. Crizotinib will be taken continuously until disease progression or unacceptable toxicity, in continuous treatment cycles of 28 days each, for a maximum of 12 cycles. Clinical response will be assessed by MRI (volumetrics, primary objective) and audiology at the end of every 3rd cycle. Subjects with volumetric tumor progression will be taken off protocol. Patients who complete 12 cycles of treatment without disease progression, but within the following 24 weeks show subsequent disease progression (defined as >20% increase in target tumor volume compared to off-treatment volume), will be eligible for re-treatment on study for up to 48 additional weeks, provided they still meet study eligibility criteria.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Oral

SUMMARY:
Subjects with Neurofibromatosis Type 2 (NF2) and progressive vestibular schwannoma (VS) will be treated with crizotinib administered orally. Crizotinib will be taken continuously until disease progression or unacceptable toxicity, in continuous treatment cycles of 28 days each, for a maximum of 12 cycles.

DETAILED DESCRIPTION:
Subjects with Neurofibromatosis Type 2 (NF2) and progressive vestibular schwannoma (VS) will be treated with crizotinib administered orally. Crizotinib will be taken continuously until disease progression or unacceptable toxicity, in continuous treatment cycles of 28 days each, for a maximum of 12 cycles. Clinical response will be assessed by MRI (volumetrics, primary objective) and audiology at the end of every 3rd cycle. Subjects with volumetric tumor progression will be taken off protocol. Patients who complete 12 cycles of treatment without disease progression, but within the following 24 weeks show subsequent disease progression (defined as >20% increase in target tumor volume compared to off-treatment volume), will be eligible for re-treatment on study for up to 48 additional weeks, provided they still meet study eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

Patients must have a confirmed diagnosis of neurofibromatosis 2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria, or by detection of a causative mutation in the NF2 gene.

The NIH criteria include presence of:

* Bilateral vestibular schwannomas, OR
* First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR
* Two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity.

The Manchester criteria include presence of:

* Bilateral vestibular schwannomas, OR First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR - Two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity OR
* Unilateral vestibular schwannoma AND any two of: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
* Multiple meningiomas (two or more) AND unilateral vestibular schwannoma OR
* Any two of: schwannoma, glioma, neurofibroma, cataract.

Patients must have progressive and measurable disease, defined as at least one VS with the following qualities:

* ≥ 0.75 ml (on volumetric analysis) that can be accurately measured by contrast-enhanced cranial MRI scan with fine cuts through the internal auditory canal (1 mm slices, no skip)
* MRI evidence of progression over the past 18 months (defined as ≥20% annualized increase in volume)

Age ≥ 6 years on day 1 of treatment.

Life expectancy of greater than 1 year.

Lansky/Karnofsky performance status ≥ 60

Organ and marrow function as defined below:

* Absolute neutrophil count ≥ 1,500/ μl
* Platelets ≥ 100,000/ μl
* Total bilirubin within ≤ 1.5 X institutional upper limit of normal
* AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
* Patients must have a creatinine clearance or radioisotope GFR ≥60ml/min/1.73 ≥60ml/min/1.73 m2 or a normal serum creatinine based on age/gender described in the table below:
* Age: 6 to < 10 years with a Maximum Serum Creatinine (mg/dL) of 1 for Male and 1 for Female
* Age: 10 to < 13 years with a Maximum Serum Creatinine (mg/dL) of 1.2 for Male and 1.2 for Female
* Age: 13 to < 16 years with a Maximum Serum Creatinine (mg/dL) of 1.5 for Male and 1.4 for Female
* Age: ≥ 16 years with a Maximum Serum Creatinine (mg/dL) of 1.7 for Male and 1.4 for Female

The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC.

Fully recovered from acute toxic effects of any prior chemotherapy, biological modifiers or radiotherapy

Any neurologic deficits must be stable for ≥1 week

Patient or parent/legal guardian must be able to provide signed informed consent and assent (as applicable for minors)

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

Patients currently receiving medical anticancer therapies or who have received medical anticancer therapies within 4 weeks of the start of study drug (including chemotherapy and molecular targeted agents), as these may interfere with the study drug

Monoclonal antibody treatment and/or agents with prolonged half-lives: At least three half-lives must have elapsed from the last dose prior to enrollment

Radiation therapy to a study target tumor within 1 year prior to enrollment, or any radiation therapy within 4 weeks prior to enrollment, as these may interfere with our ability to assess response to study drug

Prior treatment with any investigational drug within the preceding 4 weeks, as they may interfere with the study drug

Unstable or rapidly progressive disease, including patients who require glucocorticoids for symptomatic control of brain or spinal tumors, as this would represent a high risk for inability to comply with the study requirements

Use of drugs or foods that are known potent CYP3A4 inhibitors, including but not limited to ketoconazole, itraconazole, miconazole, clarithromycin, erythromycin, ritonavir, indinavir, nelfinavir, saquinavir, amprenavir, delavirdine, nefazodone, diltiazem, verapamil, and grapefruit juice, as this would interfere with study drug metabolism

Use of drugs that are known potent CYP3A4 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, tipranavir, ritonavir, and St. John's wort, as this would interfere with study drug metabolism

Use of drugs that are CYP3A4 substrates with narrow therapeutic indices, including but not limited to pimozide, aripiprazole, triazolam, dihydroergotamine, ergotamine, astemizole, cisapride, terfenadine and halofantrine, as this would interfere with study drug metabolism

Ongoing cardiac dysrhythmias of CTCAE grade ≥2, uncontrolled atrial fibrillation of any grade or prolonged QTc interval (>480 msec), as patients with these conditions would be expected to have an increased risk for cardiac toxicity related to study drug

Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

* symptomatic congestive heart failure of New York heart Association Class III or IV
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 90% or less at rest on room air
* active (acute or chronic) or uncontrolled severe infections liver disease, such as cirrhosis or severe hepatic impairment (Child-Pugh class C)

Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of crizotinib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)

Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 90 days after the last dose of study drug, as the effects of crizotinib on an unborn fetus are not known. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to administration of crizotinib.

Male patients whose sexual partner(s) are women of child bearing potential, who are not willing to use adequate contraception during the study and for 90 days after the last dose of study drug.

History of significant noncompliance to medical regimens that would jeopardize compliance with study therapy

Patients unwilling to or unable to comply with the study protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Volumetric Response Rate | Up to 48 Weeks
  estimate the best objective volumetric response rates (i.e. maximum tumor shrinkage) to crizotinib in NF2 patients with VS during up to 12 cycles (48 weeks) of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Girish Dhall, MD, Study Director — University of Alabama at Birmingham; Matthias A Karajannis, MD, MS, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (15):
- United States (15):
  - The University of Alabama at Birmingham (Site 700), Birmingham, Alabama
  - Univ of California @ Los Angeles (Site 325), Los Angeles, California
  - Children's National Medical Center (Site 775), Washington D.C., District of Columbia
  - Children's HealthCare of Atlanta (Site 950), Atlanta, Georgia
  - Lurie Childrens Hospital of Chicago (Site 350), Chicago, Illinois
  - University of Chicago (Site 850), Chicago, Illinois
  - Indiana University (Site 400), Indianapolis, Indiana
  - Johns Hopkins University (Site 250), Baltimore, Maryland
  - Children's Hospital Boston (Site 725), Boston, Massachusetts
  - Washington University - St. Louis (Site 900), St Louis, Missouri
  - New York University Medical Center (Site 200), New York, New York
  - Memorial Sloan Kettering Cancer Center (Site 210), New York, New York
  - Cincinnati Children's Hospital Medical Center (Site 800), Cincinnati, Ohio
  - Children's Hospital of Philadelphia (Site 750), Philadelphia, Pennsylvania
  - Childrens Medical Center - Univ. of Texas SW (Site 917), Dallas, Texas

IPD SHARING:
Plan to Share IPD: No